CLINICAL TRIAL: NCT04276376
Title: A Multicenter, Open Label, Phase II Basket Trial Exploring the Efficacy and Safety of the Combination of Rucaparib (PARP Inhibitor) and Atezolizumab (Anti-PD-L1 Antibody) in Patients With DNA Repair-deficient or Platinum-sensitive Solid Tumors
Brief Title: Efficacy and Safety of the Combination of Rucaparib (PARP Inhibitor) and Atezolizumab (Anti-PD-L1 Antibody) in Patients With DNA Repair-deficient or Platinum-sensitive Solid Tumors
Acronym: ARIANES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Bankruptcy of partner: Clovis
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001744-62; 2018/2727 (Other: CSET number)
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — atezolizumab; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1A-D (Experimental): Molecularly selected cohorts that harbor DNA repair deficiency, defined as bi-allelic loss-of-function alteration (mutation and/or deletion) in at least one of the following genes: ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK2, PALB2, RAD51C, RAD51D, FANCA, NBN, RAD51, RAD54L.
  1.A - Non-Small Cell Lung Cancer
  1.B - Urothelial Bladder Cancer
  1.C - metastatic Castration Resistant Prostate Cancer
  1.D - others: any histology, excepted breast cancer or serous ovarian cancer
  Interventions: Drug: Atezolizumab; Drug: Rucaparib
- Cohort 2A-C (Experimental): Platinum-sensitive disease 2.A - Non-Small Cell Lung Cancer 2.B - Urothelial Bladder Cancer 2.C - Gastric or gastro-esophageal junction adenocarcinoma
  Interventions: Drug: Atezolizumab; Drug: Rucaparib
- Cohort 3 (Experimental): Metastatic Castration Resistant Prostate Cancer (mCRPC)
  Interventions: Drug: Atezolizumab; Drug: Rucaparib
- Cohort 4 (Experimental): Clear Cell Renal Cell Carcinoma
  Interventions: Drug: Atezolizumab; Drug: Rucaparib

INTERVENTIONS:
Drug: Atezolizumab — Fc-engineered, humanized, Ig G1 monoclonal antibody against PDL-1 1200mg q3w
Drug: Rucaparib — Inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) 600mg BID

SUMMARY:
The primary objective of the trial is to evaluate the antitumor activity of atezolizumab and rucaparib in patients with selected advanced solid tumors as measured by the Overall Response Rate

ELIGIBILITY:
INCLUSION CRITERIA

1. Signed informed consent form.
2. Age ≥ 18 years.
3. Patients must have histologically or cytologically confirmed progressive metastatic or recurrent solid tumor (as defined below for each tumor type). Diagnosis must be stated in a pathology report and confirmed by the investigator.
4. To be enrolled in this study, only the tumor types and settings described below are allowed:

   4.1 - Cohorts 1 A-D: DNA repair deficiency, defined as bi-allelic loss-of-function alteration (mutation and/or deletion) in at least one of the following genes: ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK2, PALB2, RAD51C, RAD51D, FANCA, NBN, RAD51, RAD54L.

   4.1.1 - Cohort 1A: Non Small Cell Lung Cancer 4.1.2 - Cohort 1B: Urothelial Bladder Cancer 4.1.3 - Cohort 1C: metastatic Castration Resistant Prostate Cancer (mCRPC) 4.1.4 - Cohort 1D: Others 4.2 - Cohorts 2A-C: Platinum-sensitive disease 4.2.1 - Cohort 2A: Non Small Cell Lung Cancer 4.2.2 - Cohort 2B: Urothelial Bladder Cancer 4.2.3 - Cohort 2C: Gastric or gastro-esophageal junction adenocarcinoma 4.3 - Cohort 3: Metastatic Castration Resistant Prostate Cancer (mCRPC) 4.4 - Cohort 4: Clear cell Renal Cell Carcinoma
5. Representative archival formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (preferred) or 20 freshly cut and unstained slides, with an associated pathology report, for ancillary studies and central testing, is mandatory for all cohorts. In all cases, recovery of the most recent tumor block or biopsy is encouraged and tumor tissue has to date back from less than 3 years ago (less than 6 years for cohort 4). Cohorts 1 and 2: if tumor tissue is more than 3 years old, a fresh tumor biopsy is mandatory. Cohort 4: if tumor tissue is more than 6 years old, a fresh tumor biopsy is mandatory.

   * Specificities for Cohorts 1A-D:
   * For patients with DNA repair gene mutation already identified by local testing, mutational testing must have been done less than one year prior to inclusion in the trial (i.e. signing of informed consent). Tumor block should correspond to the one that has been used for the original testing. If more recent blocks are available, these should be provided for ancillary studies, and the presence of the mutation of interest should be confirmed on these.
   * If no archival tissue is available or if tumor tissue is more than 3 years old, feasibility of a fresh tumor biopsy at baseline (C0D1 pre-dose) should be ensured and mutation confirmed on that tissue for cohorts 1A, 1B and 1D. Only tissue from core needle, punch or excisional biopsy sample collection will be accepted. Other methods such as fine-needle aspiration, brushing, bone tissue or lavage samples are not acceptable.
   * Bone biopsies are allowed for mCRPC (cohort 1C), if sufficient tumor cellularity can be achieved.
   * Specificity for cohort 3:
   * If no archival tumor biopsy is available, a new fresh biopsy should be done prior to treatment start (C0D1 pre-dose) whenever feasible; otherwise, any archival tumor tissue will be accepted.
   * Core or excisional biopsy from soft tissue or a bone biopsy is required from a site not previously irradiated (samples from tumors progressing in a prior site of radiation are allowed; other exceptions may be considered after Sponsor consultation).
6. Measurable disease, defined as:

   * For the non-prostate cohorts: At least one lesion, not previously irradiated, measurable according to RECIST v1.1 as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and suitable for repeated assessment.
   * For prostate cohorts: At least one lesion, not previously irradiated, measurable according to RECIST v1.1 and / or bone scan measurable disease (Cf inclusion criteria 4) and / or measurable disease according to Prostate Cancer Working Group Criteria 3 (PCWG3)
7. Agreement of the patient to sign the genetic analysis consent form for access to plasma samples for ctDNA analysis.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration from registration date.
9. Estimated life expectancy of greater than 12 weeks.
10. Adequate hematologic and organ function, defined by the following laboratory results obtained within 3 days prior to the first study treatment (Cycle 0 Day 1):

    * Absolute neutrophil count (ANC) ≥ 1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks before cycle 0 day 1).
    * Platelet count ≥ 100.000/μL (without transfusion within 2 weeks before Cycle 0 Day 1).
    * Hemoglobin ≥ 9g/dL (patients may be transfused or receive erythropoietic treatment to meet this criterion).
    * Total bilirubin ≤ 1.5 ULN (subjects with documented/suspected Gilbert's disease or liver metastases may be enrolled with bilirubin ≤ 3 × ULN).
    * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit (ULN) or ≤ 5 × ULN in case of liver metastases.
    * Albumin ≥ 28g/L.
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 40mL/min .
    * International normalized ratio and activated partial thromboplastin time ≤ 1.5 x ULN. This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular weight heparin or warfarin) should be on stable dose.
11. Women of childbearing potential must have a negative serum β-HCG pregnancy test within 7 days prior to the administration of the first study treatment
12. Sexually active women of childbearing potential must agree to use a highly effective method of contraception << supplemented by a barrier method >>, or to abstain from sexual activity during the study and for at least 6 months after the last study treatment administration.
13. Sexually active males patients must agree to use condom during the study and for at least 6 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception.

    A woman is considered of childbearing potential following menarche and until becoming post-menopausal (≥ 12 months of non-therapy-induced amenorrhea) unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral oophorectomy and bilateral salpingectomy.

    A highly effective birth control method is a one which can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include: combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation; progestogen-only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence during the entire period of risk associated with study treatment. To prevent the risk of interaction between the study drug and hormonal contraceptives, hormonal contraceptives should be supplemented with a barrier method (preferably male condom). Following methods are considered as unacceptable methods (non-exhaustive list): periodic abstinence (calendar, symptothermal, post-ovulation methods) and withdrawal (coitus interruptus).
14. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
15. Patient should be able and willing to comply with study visits and procedures as per protocol.
16. Patients must be affiliated to a social security system or beneficiary of an equivalent system.

NON-INCLUSION CRITERIA

Any of the following would exclude the subject from participation in the study:

1. Participation in another clinical study with an investigational product during the last 4 weeks (excepting non-interventional clinical studies) and while on study treatment.
2. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy (excepted androgen deprivation therapy by LHRH agonists for prostate cancer patients), targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug, or five half lives of the previous agent, whichever is the shorter.
3. Prior radiation therapy within 2 weeks prior to Cycle 0 Day 1.
4. History of another primary malignancy within 5 years prior to Cycle 0 Day 1 except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease (eg, carcinoma in situ of the cervix, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
5. Treatment with systemic corticosteroids or other immunosuppressive medications within 2 weeks prior to Cycle 0 Day 1, or anticipated requirements for systemic immunosuppressive medications during the trial:

   . The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids for patients with orthostatic hypotension, low-dose supplemental corticosteroids for adrenocortical insufficiency and topical steroids for cutaneous diseases are allowed.
6. Acute toxicities from previous therapies that have not resolved to Grade ≤ 1, with the exception of alopecia.
7. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1.
8. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
9. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation.
10. History of autoimmune/immune mediated inflammatory disease, including but not limited to colitis, pneumonitis, hepatitis, hypophysitis, nephritis, hyperthyroidism, systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, vasculitis, or glomerulonephritis (see Appendix 2) excepted stable hypothyroidism or stable Type 1 diabetes mellitus.
11. Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis).
12. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan - History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
13. History of allogeneic organ transplant or prior bone marrow transplantation of double umbilical cord blood transplantation.
14. Uncontrolled intercurrent illness including, but not limited to:

    * ongoing or active infection or severe infection requiring hospitalization or IV antibiotics within 2 weeks of starting treatment (with the exception of prophylactic antibiotics).
    * symptomatic congestive heart failure > NYHA II, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, pericardial effusion.
    * active peptic ulcer disease or gastritis.
    * active bleeding diatheses.
15. Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
16. Patients with known left ventricular ejection fraction (LVEF) < 40%; patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable cardiologic treatment.
17. Known positive test for HIV.
18. Patients with active hepatitis B (defined as positive HBsAg test at screening) or hepatitis C (HCV). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen anti-HBc) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
19. Active tuberculosis.
20. Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. - Influenza vaccination should be given during influenza season only (example: approximately October to March in the Northern Hemisphere). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study treatment or within 5 months after the last dose of atezolizumab.
21. Major surgical procedure within 28 days prior to Cycle 0 Day 1 or anticipation of need for a major surgical procedure during the course of the study.
22. Uncontrolled tumor-related pain: patients requiring pain medication must be on a stable regimen at study entry and symptomatic lesions amenable to palliative radiotherapy should be treated prior to enrollment.
23. Uncontrolled effusion (pleural, pericardial or ascites) requiring recurrent drainage procedures (once a month or more frequently); patients with indwelling catheters (e.g. PleurX) are allowed.
24. Uncontrolled hypercalcemia (>1.5mmol/L ionized calcium or Ca > 12mg/dL or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
25. Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history or clinically significant hypercalcemia are eligible
26. History of leptomeningeal disease

    * Symptomatic CNS metastasis or uncontrolled CNS metastasis, requiring increasing doses of steroids or stable dose of steroids > 10mg prednisone qd.
    * Spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to Cycle 0 Day 1.
27. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
28. Previous treatment with PARP inhibitors.
29. Concomitant use of strong inhibitors or inducers of CYP3A4 (See Appendix 3).
30. Treatment with systemic immunostimulatory agents (e.g. INF-a and IL-2) within 4 weeks prior to Cycle 0 Day 1.
31. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study result.
32. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No